CLINICAL TRIAL: NCT05318365
Title: Bladder and Bowel Dysfunction in Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BBD_Children
Record Dates: First submitted 2022-03-30; First posted 2022-04-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Bladder and Bowel Dysfunction
Keywords: Dysfunctional Elimination Syndrome; Urinary Incontinence in Children; Functional constipation in Children; Gut Microbiome; Urine Microbiome
MeSH Terms: conditions — Intestinal Diseases | interventions — polyethylene glycol 3350; Magnesium Oxide; picosulfate sodium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment of constipation and/or faecal incontinence (Active Comparator): Medical treatment of bowel symptoms in accordance with the guidelines of The European Society for Paediatric Gastroenterology, Hepatology and Nutrition
  Interventions: Drug: Polyethylene Glycol 3350
- Treatment of constipation and/or faecal incontinence combined with urotherapy (Active Comparator): Medical treatment of bowel symptoms in accordance with the guidelines of The European Society for Paediatric Gastroenterology, Hepatology and Nutrition combined with standard urotherapy in accordance with International Children's Continence Society (ICCS)
  Interventions: Drug: Polyethylene Glycol 3350; Behavioral: Urotherapy

INTERVENTIONS:
Drug: Polyethylene Glycol 3350 — PEG3350, klysma, laxoberal and magnesia will be administered in accordance with actual guidelines for treatment of constipation in children
  Other Names: Magnesia; Laxoberal; Glyoktylklysma
Behavioral: Urotherapy — Information and demystification of the disorder along with behavioural modification such as timed voiding, proper voiding posture, avoidance of holding manoeuvers and balanced fluid intake
  Arms: Treatment of constipation and/or faecal incontinence combined with urotherapy

SUMMARY:
Background:

Bladder and bowel dysfunction (BBD) is characterized by lower urinary tract symptoms accompanied by bowel complaints. BBD is a common condition in childhood. The present treatment strategy for BBD is a step-wise approach starting with management of bowel symptoms before initiation of standard urotherapy and further medical treatment of LUTS symptoms. This is, however, based on clinical experience and few retrospective, non-randomized studies and high-level evidence of the succession of the elements in treatment of BBD children is missing.

Our microbiome, and its role in health and disease, has gained increased focus during the past years. Studies suggest the urine and gut microbiome to be critical for maintenance of a well-functioning bladder- and bowel system. The microbiome in children is only sparsely investigated and its role in BBD is to the investigator's knowledge still unexplored.

Study 1:

Aim: To investigate if combination therapy is more effective in treating urinary incontinence in BBD children.

Materials and methods: A prospective randomized multicentre study on children with BBD (n=100) between 5-14 years and 9 months old. They are randomized to: 1) Medical treatment of bowel symptoms (n=50) or 2) Medical treatment of bowel symptoms combined with standard urotherapy.

The effect of treatment will be evaluated after 3 months. Primary endpoint: Resolution of incontinence after treatment. Secondary endpoint: Improved quality of life after successful treatment of urinary incontinence.

Study 2:

Aim: To investigate the urofecal microbiome in children with BBD

Materials and methods:

1. A cohort study to investigate, whether the urofecal microbiome can predict response to treatment and whether it changes during treatment period
2. A case control study to investigate whether the urofecal microbiome is different in children with BBD and recurrent UTI 's and children with BBD without recurrent UTI 's.

The study population consists of children with BBD included in study 1. A urine-, stool sample and a perineum swab will be collected from all participants before and after treatment. Bacterial DNA will be extracted and the microbiome will be determined.

Perspectives:

BBD is a common condition in childhood. It is associated with a considerable psychological burden and a risk of more severe physical complications.

The studies will provide basic knowledge about characteristics of the BBD patients and contribute new information about the optimal treatment of BBD children.

DETAILED DESCRIPTION:
Background Bladder and bowel dysfunction (BBD) is characterised by lower urinary tract symptoms (LUTS) accompanied by bowel complaints, primarily functional constipation and/or faecal incontinence. To standardise the terminology used for BBD, LUTS symptoms related to the disease have been defined by International Children's Continence Society (ICCS).

The prevalence of BBD is probably underestimated but studies suggest BBD to be present in up to 20 % of school children and to represent up to 40% of paediatric urology consults.

Embryological, anatomical and functional interactions between the rectum and urinary bladder are well known. Bladder and bowel are anatomically closely related and share innervation from the parasympathetic S2-S4 and sympathetic L1-L3 nerve roots.

Research on successful treatment of BBD is sparse, with only few retrospective, non-randomized studies, documenting that treatment of defecation problems in children with BBD enhances successful management of lower urinary tract disturbances such as daytime urinary incontinence (DUI), enuresis and urinary tract infections (UTI's). Based on this knowledge and clinical experience, the present treatment strategy for children with BBD is a step-wise approach starting with management of bowel symptoms before initiation of standard urotherapy and further medical treatment of LUTS symptoms. Standard urotherapy encompasses information and demystification of the disorder along with behavioural modification such as timed voiding, proper voiding posture, avoidance of holding manoeuvers and balanced fluid intake. Standard urotherapy is well-established as first-line treatment for children with LUTS. However, high-level evidence of the succession of the elements in treatment of BBD children is missing.

BBD is commonly associated with vesicoureteral reflux (VUR) and recurrent UTI's, which may lead to renal scarring , kidney failure and hypertension. It is a potential cause of significant physical and psychosocial burden for children and families. Therefore, optimization of treatment is critical to avoid secondary comorbidities.

Our microbiome, and its role in health and disease, has gained increased focus during the past few years.

Studies suggest the urine and gut microbiome to be critical for maintenance of a well-functioning bladder- and bowel system.

Dysbiosis is defined by the presence of unbalanced and disease-promoting composition of the microbiome. It is well-established that dysbiosis is associated with constipation in children and the condition is suspected to be involved in urological disorders such as overactive bladder, urge, incontinence and recurrent UTI's in adults. However, the composition of the urine microbiome in children is only sparsely investigated and its role in BBD and childhood UTI's is to the investigator's knowledge still unexplored.

Study 1: Does successful treatment of bowel symptoms resolve urinary incontinence in children with BBD? Aim and hypothesis Aim: To investigate if effective treatment of bowel problems resolves urinary incontinence in BBD children.

The hypothesis of the investigators is:

1. Treatment of bowel symptoms resolves urinary incontinence in BBD children.
2. It is more effective to initiate urotherapy from the beginning in combination with treatment of bowel symptoms instead of the present regime where bowel symptoms are managed before urotherapy is started.
3. Succesful treatment of urinary incontinence in children with BBD improves their quality of life.

1.2 Materials and methods A prospective multicentre randomised study on children with BBD referred to the Pediatric Incontinence and Gastroenterology outpatient clinics at the Department of Pediatrics, Aarhus University Hospital, Aalborg University Hospital and Regional Hospital Goedstrup.

Children (n=100) between 5-14 years and 9 months diagnosed with BBD at their first visit to the outpatient clinic will be included if they meet in- and exclusion criteria.

The included children will be randomised to one of the following treatments:

1. Medical treatment of bowel symptoms in accordance with the guidelines of The European Society for Paediatric Gastroenterology, Hepatology and Nutrition (ESPGHAN) (n=50)
2. Medical treatment of bowel symptoms in accordance with the ESPGHAN guidelines combined with standard urotherapy (n=50)

At first visit to the outpatient clinic, enrolled children will undergo physical examination including neurological examination. Data on medical history will be collected including number of and time for UTI's. Participants will be asked to fill in a 48-hour flow-volume chart and in case of enuresis nocturna the chart will also include registration for 7 nights. Participants will also fill in "Toerfisk" which is a validated tool to monitor severity of urinary incontinence. Routine uroflowmetry will be performed for further evaluation of lower urinary symptoms. A urine sample will be collected for diagnosing on-going UTI and for microbiome analysis in study 3. The children will be screened for constipation in accordance with the ROME IV criteria. Rectal examination will be performed or transrectal diameter will be evaluated with point-of-care ultrasound. Stool sample and perineum swab will be collected for microbiome analysis.

The psychological burden from the children´s BBD condition will be evaluated by PinQ, a validated questionnaire used for assessment of quality of life according to the incontinence issue of the patients.

All participants will be informed about bladder and bowel function in order to demystify the disorder. Daily defecation will be induced by reconditioning to normal bowel habits through timed toilet sitting and daily administration of laxatives (e.g. PEG3350) in relevant dosage according to the ESPGHAN guidelines.

Participants randomized to combined medical treatment for bowel symptoms and urotherapy will be instructed in urotherapy in accordance with earlier description.

After 1 month of treatment the participants will be contacted by telephone to ensure compliance and for adjustment of laxative dose depending on the bowel symptoms.

The second visit in the outpatient clinic will be after 3 months of treatment. Before the consultation, the participants will be asked to fill in a second flow-volume chart as well as "Toerfisk" and PinQ questionnaires. Uroflowmetry will be repeated and a second urine sample will be collected for stix, culturing and microbiome analysis. Bowel symptoms will be evaluated using ROME IV, rectal examination and transrectal diameter and a second stool sample and perineum swab will be collected for microbiome analysis for study 3.

Data storage Data will be entered into RedCap, which is a secure web platform for building and managing online databases.

Power estimation The sample size (n=100) was calculated for each group to achieve a power of 80% for detecting a difference in proportions of 0.30 between the two groups (test - reference group) at a two sided p-value of 0.05.

Study 2: Urine, perineal and gut microbiome in children with BBD before and after treatment Aim and hypothesis To investigate the urine, perineal and gut microbiome in children with BBD before and after treatment.

The hypothesis of the investigators is that

1. Response to treatment can be predicted by the composition of the urine, perineal and gut microbiome in children with BBD.
2. The composition of the urine, perineal and gut microbiome is different in BBD children with recurrent UTI's compared to BBD children without recurrent UTI's.
3. The urine, perineal and gut microbiome in children with BBD will change when bladder and bowel symptoms successfully treated.

Materials and methods

The study is a multicentre study consisting of two elements:

1. a cohort study to investigate, whether the urine, perineal and gut microbiome can predict response to treatment and whether it changes during treatment period
2. a case control study to investigate whether the urine, perineal and gut microbiome is different in children with BBD and recurrent UTI 's and children with BBD without recurrent UTI 's.

The study population consists of children with BBD included in study 1.

Collection and analysis of samples A urine-, stool sample and a perineum swab will be collected from all participants before initiation of treatment and after 3 months of treatment as described in study 1. Bacterial DNA will be extracted and the microbiome will be determined.

Data storage Biological material will be pseudonymised and stored in a -80 degree fridge until analysis is performed.

Statistical analysis for all 3 studies Distribution and variance will be analysed by QQ plot, Shapiro-Wilks test and Bartletts test. Microbiota alpha-diversity will be addressed by ASV richness, Faith's phylogenetic diversity, Shannon diversity index, and Pielou's evenness index. Beta-diversity analysis will include principal coordinate analysis (PCoA) using Bray-Curtis dissimilarity, weighted and unweighted UniFrac. Parametric data will be compared using Student's t-test or one-way ANOVA and Tukey´s post hoc test, while non-parametric data will be compared with Kruskal-Wallis test or Mann-Whitney U-test. Chi Squared test will be used for proportions. Level of significance will be as following *: p <0.05, **: p<0.01 and ***: p<0.001.

Ethics The studies will be conducted in accordance with the Declaration of Helsinki. All side effects will be handled in accordance with the actual legislation. No risk or unknown side effects are expected to urotherapy or medical treatment of bowel symptoms. No risk, side effects or discomfort is expected from collection of urine, stool and perineum samples or from uroflowmetry or transabdominal ultrasound.

Perspectives BBD is a common condition in childhood. It is associated with a considerable psychological burden and a risk of more severe physical complications.

The term BBD is recently defined and therefore only sparsely investigated. The studies will provide basic knowledge about characteristics of the BBD patients and contribute new information about the optimal treatment of BBD children.

ELIGIBILITY:
Inclusion Criteria:

* Age 5-14 years and 9 months at time of inclusion
* Diagnosed with urinary incontinence and/or enuresis nocturna defined by the ICCS criteria
* Diagnosed with constipation and/or faecal incontinence defined by the ROME IV criteria
* Normal clinical examination
* Parents/guardian can understand the written and spoken information
* Informed assent to participation from both parents/guardian

Exclusion Criteria:

* Neuropathic or anatomical abnormalities in the urinary tract or gastrointestinal canal
* Earlier surgical intervention of the urinary tract (except circumcision)
* Neurological illness or earlier cerebral surgical intervention
* On-going urinary tract infection
* On-going treatment with anticholinergics and/or β3-adenoceptoragonist
* On-going treatment with laxatives in correct dosage (PEG3350 1-2 g/kg/day)
* Inflammatory bowel disease
* Other disorder affection bladder or bowel function
* For Study 2 (microbiome): Systemic antibiotics within the past 3 months

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with reduction in weekly episodes of urinary incontinence | Evaluation after 3 months of treatment
  No-response: <50% reduction, Partial response: 50 to 99% reduction, Complete response: 100% reduction.

SECONDARY OUTCOMES:
Number of participants with a change in quality of life after succesful treatment of urinary incontinence | Evaluation after 3 months of treatment
  Tool: PinQ Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Sofie Axelgaard, MD, Study Chair — Department of Childhood and Adolescent Medicine, Regional Hospital Goedstrup; Soeren Hagstroem, Professor, MD, Principal Investigator — Department of Childhood and Adolescent Medicine, Aalborg University Hospital; Luise Borch, MD, PhD, Study Director — Department of Childhood and Adolescent Medicine, Regional Hospital Goedstrup; Konstantinos Kamperis, MD, PhD, Study Director — Department of Childhood and Adolescent Medicine, Aarhus University Hospital
Locations (3):
- Denmark (3):
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - Goedstrup Regional Hospital, Herning

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Conway PH, Cnaan A, Zaoutis T, Henry BV, Grundmeier RW, Keren R. Recurrent urinary tract infections in children: risk factors and association with prophylactic antimicrobials. JAMA. 2007 Jul 11;298(2):179-86. doi: 10.1001/jama.298.2.179. PMID 17622599
- [Background] Aguiar LM, Franco I. Bladder Bowel Dysfunction. Urol Clin North Am. 2018 Nov;45(4):633-640. doi: 10.1016/j.ucl.2018.06.010. Epub 2018 Sep 7. PMID 30316317
- [Background] Shaikh N, Hoberman A, Wise B, Kurs-Lasky M, Kearney D, Naylor S, Haralam MA, Colborn DK, Docimo SG. Dysfunctional elimination syndrome: is it related to urinary tract infection or vesicoureteral reflux diagnosed early in life? Pediatrics. 2003 Nov;112(5):1134-7. doi: 10.1542/peds.112.5.1134. PMID 14595058
- [Background] Dos Santos J, Varghese A, Koyle M. Recommendations for the management of bladder bowel dysfunction in children. Pediatr Therapeut, 2014;4:1.
- [Background] Halachmi S, Farhat WA. Interactions of constipation, dysfunctional elimination syndrome, and vesicoureteral reflux. Adv Urol. 2008;2008:828275. doi: 10.1155/2008/828275. PMID 18604297
- [Background] Kaplan SA, Dmochowski R, Cash BD, Kopp ZS, Berriman SJ, Khullar V. Systematic review of the relationship between bladder and bowel function: implications for patient management. Int J Clin Pract. 2013 Mar;67(3):205-16. doi: 10.1111/ijcp.12028. PMID 23409689
- [Background] Koff SA, Wagner TT, Jayanthi VR. The relationship among dysfunctional elimination syndromes, primary vesicoureteral reflux and urinary tract infections in children. J Urol. 1998 Sep;160(3 Pt 2):1019-22. doi: 10.1097/00005392-199809020-00014. PMID 9719268
- [Background] Chase JW, Homsy Y, Siggaard C, Sit F, Bower WF. Functional constipation in children. J Urol. 2004 Jun;171(6 Pt 2):2641-3. doi: 10.1097/01.ju.0000109743.12526.42. PMID 15118440
- [Background] Erickson BA, Austin JC, Cooper CS, Boyt MA. Polyethylene glycol 3350 for constipation in children with dysfunctional elimination. J Urol. 2003 Oct;170(4 Pt 2):1518-20. doi: 10.1097/01.ju.0000083730.70185.75. PMID 14501649
- [Background] Borch L, Hagstroem S, Bower WF, Siggaard Rittig C, Rittig S. Bladder and bowel dysfunction and the resolution of urinary incontinence with successful management of bowel symptoms in children. Acta Paediatr. 2013 May;102(5):e215-20. doi: 10.1111/apa.12158. Epub 2013 Feb 11. PMID 23368903
- [Background] Hoebeke P, Bower W, Combs A, De Jong T, Yang S. Diagnostic evaluation of children with daytime incontinence. J Urol. 2010 Feb;183(2):699-703. doi: 10.1016/j.juro.2009.10.038. Epub 2009 Dec 21. PMID 20022025
- [Background] Loening-Baucke V. Urinary incontinence and urinary tract infection and their resolution with treatment of chronic constipation of childhood. Pediatrics. 1997 Aug;100(2 Pt 1):228-32. doi: 10.1542/peds.100.2.228. PMID 9240804
- [Background] Hagstroem S, Rittig N, Kamperis K, Mikkelsen MM, Rittig S, Djurhuus JC. Treatment outcome of day-time urinary incontinence in children. Scand J Urol Nephrol. 2008;42(6):528-33. doi: 10.1080/00365590802098367. PMID 18609267
- [Background] Mulders MM, Cobussen-Boekhorst H, de Gier RP, Feitz WF, Kortmann BB. Urotherapy in children: quantitative measurements of daytime urinary incontinence before and after treatment according to the new definitions of the International Children's Continence Society. J Pediatr Urol. 2011 Apr;7(2):213-8. doi: 10.1016/j.jpurol.2010.03.010. Epub 2010 Jun 11. PMID 20541978
- [Background] Keren R, Shaikh N, Pohl H, Gravens-Mueller L, Ivanova A, Zaoutis L, Patel M, deBerardinis R, Parker A, Bhatnagar S, Haralam MA, Pope M, Kearney D, Sprague B, Barrera R, Viteri B, Egigueron M, Shah N, Hoberman A. Risk Factors for Recurrent Urinary Tract Infection and Renal Scarring. Pediatrics. 2015 Jul;136(1):e13-21. doi: 10.1542/peds.2015-0409. Epub 2015 Jun 8. PMID 26055855
- [Background] Patzer L, Seeman T, Luck C, Wuhl E, Janda J, Misselwitz J. Day- and night-time blood pressure elevation in children with higher grades of renal scarring. J Pediatr. 2003 Feb;142(2):117-22. doi: 10.1067/mpd.2003.13. PMID 12584530
- [Background] Bower WF. Self-reported effect of childhood incontinence on quality of life. J Wound Ostomy Continence Nurs. 2008 Nov-Dec;35(6):617-21. doi: 10.1097/01.WON.0000341476.71685.78. PMID 19018203
- [Background] Equit M, Hill J, Hubner A, von Gontard A. Health-related quality of life and treatment effects on children with functional incontinence, and their parents. J Pediatr Urol. 2014 Oct;10(5):922-8. doi: 10.1016/j.jpurol.2014.03.002. Epub 2014 Mar 26. PMID 24726201
- [Background] Whiteside SA, Razvi H, Dave S, Reid G, Burton JP. The microbiome of the urinary tract--a role beyond infection. Nat Rev Urol. 2015 Feb;12(2):81-90. doi: 10.1038/nrurol.2014.361. Epub 2015 Jan 20. PMID 25600098
- [Background] Nishida A, Inoue R, Inatomi O, Bamba S, Naito Y, Andoh A. Gut microbiota in the pathogenesis of inflammatory bowel disease. Clin J Gastroenterol. 2018 Feb;11(1):1-10. doi: 10.1007/s12328-017-0813-5. Epub 2017 Dec 29. PMID 29285689
- [Background] de Moraes JG, Motta ME, Beltrao MF, Salviano TL, da Silva GA. Fecal Microbiota and Diet of Children with Chronic Constipation. Int J Pediatr. 2016;2016:6787269. doi: 10.1155/2016/6787269. Epub 2016 Jun 23. PMID 27418934
- [Background] Petersen C, Round JL. Defining dysbiosis and its influence on host immunity and disease. Cell Microbiol. 2014 Jul;16(7):1024-33. doi: 10.1111/cmi.12308. Epub 2014 Jun 2. PMID 24798552
- [Background] Pearce MM, Hilt EE, Rosenfeld AB, Zilliox MJ, Thomas-White K, Fok C, Kliethermes S, Schreckenberger PC, Brubaker L, Gai X, Wolfe AJ. The female urinary microbiome: a comparison of women with and without urgency urinary incontinence. mBio. 2014 Jul 8;5(4):e01283-14. doi: 10.1128/mBio.01283-14. PMID 25006228
- [Background] Jung C, Brubaker L. The etiology and management of recurrent urinary tract infections in postmenopausal women. Climacteric. 2019 Jun;22(3):242-249. doi: 10.1080/13697137.2018.1551871. Epub 2019 Jan 9. PMID 30624087
- [Background] Kinneman L, Zhu W, Wong WSW, Clemency N, Provenzano M, Vilboux T, Jane't K, Seo-Mayer P, Levorson R, Kou M, Ascher D, Niederhuber JE, Hourigan SK. Assessment of the Urinary Microbiome in Children Younger Than 48 Months. Pediatr Infect Dis J. 2020 Jul;39(7):565-570. doi: 10.1097/INF.0000000000002622. PMID 32091499
- [Background] Kassiri B, Shrestha E, Kasprenski M, Antonescu C, Florea LD, Sfanos KS, Wang MH. A Prospective Study of the Urinary and Gastrointestinal Microbiome in Prepubertal Males. Urology. 2019 Sep;131:204-210. doi: 10.1016/j.urology.2019.05.031. Epub 2019 Jun 10. PMID 31195012
- [Background] Levy EI, Lemmens R, Vandenplas Y, Devreker T. Functional constipation in children: challenges and solutions. Pediatric Health Med Ther. 2017 Mar 9;8:19-27. doi: 10.2147/PHMT.S110940. eCollection 2017. PMID 29388621